CLINICAL TRIAL: NCT05877612
Title: Observational, Prospective, Monocentric Study Aimed at Studying the Efficacy of Spinal Cord Stimulation in Burst Mode in the Treatment of Complex Regional Pain Syndromes (CRPS) Type 1 of the Upper Limbs Evaluation Protocol by Quantitative and Qualitative Method
Brief Title: Efficacy of Spinal Cord Stimulation in Burst Mode in the Treatment of Complex Regional Pain Syndromes Type 1 of the Upper Limbs
Acronym: STIMBURST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Elsan (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A00638-37
Record Dates: First submitted 2023-05-05; First posted 2023-05-26 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Complex Regional Pain Syndrome Type I
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Burst stimulation: Patients treated by Spinal Cord Stimulation in Burst Mode for their Complex Regional Pain Syndromes (CRPS) Type 1 of the Upper Limbs
  Interventions: Device: Implantable spinal cord stimulator

INTERVENTIONS:
Device: Implantable spinal cord stimulator — Spinal cord stimulation is possible thanks to implantable spinal cord neurostimulators. These are medical devices, which include a stimulation electrode and an implantable box, designed to deliver electrical stimulation for pain relief. The electrode is implanted in the epidural space in order to stimulate the posterior cords of the spinal cord through the dura mater, at the dorsal or cervical level.

SUMMARY:
In this study, it is the procedure of spinal cord stimulation in Burst mode, its results and the experience of the patients that are evaluated.

DETAILED DESCRIPTION:
There is 1 "classic" spinal cord stimulation setting that can be problematic in the case of cervical spinal cord stimulation because neck movements tend to trigger paresthesias. It is therefore possible, in a certain number of cases, that these side effects prevent the treatment from being effective. Thus, the development of new modes of spinal cord stimulation, mainly aiming at eliminating these side effects, has proven to be particularly interesting.

There are 3 new modes of stimulation: high frequency stimulation which uses very short pulse durations and a stimulation frequency of the order of 1000 Hz, high density stimulation which uses long duration pulses and an intermediate stimulation frequency, and "Burst" stimulation which uses stimulation trains repeated 40 times per second.

The Burst stimulation mode preferentially activates pathways in the medial part of the pain matrix, leading mainly to the cingulate cortex involved in modulating the affective, emotional and attentional side of pain. This result should theoretically be felt positively by the patient and his entourage, and the benefit should persist, or even improve with time, contrary to what is often observed with other stimulation modes.

In addition, the Burst mode consumes little energy, theoretically less than conventional stimulation. It is therefore not necessary to use rechargeable stimulators, which provides greater comfort for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years of age
* Patient with CRPS of at least one upper limb
* Patient affiliated to a Social Security plan
* Patient who has signed and dated the no-objection form
* Patient with the cognitive ability to understand the treatment and complete the questionnaires
* Patient who can be followed for a minimum of 1 year

Exclusion Criteria:

* Patient with an uncontrolled infection
* Pregnant or breastfeeding patient
* Patient who has already undergone treatment by spinal cord stimulation
* Patient with a contraindication to the percutaneous technique (cervical spine surgery, infection...)
* Patient who cannot be followed regularly for psychological, social, family or geographical reasons
* Protected participant: adult under guardianship, curatorship or other legal protection, deprived of freedom by judicial or administrative decision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Complex Regional Pain Syndromes (CRPS) Type 1 of the Upper Limbs, eligible for implantation of a medullary stimulator
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pain assessment at 3 months after implant | 3 months
  The analgesic outcome of spinal cord stimulation will be assessed by comparing the preoperative visual analogue pain scales (VAS) (ranging from 0: "No pain" to 100: "Maximum pain imaginable") to those performed at the 3rd month visit (3 months). Patients with a VAS score of 50% or more improvement will be considered "improved". The VAS value retained corresponds to the average of 3 values taken during the day (morning, noon and evening).

SECONDARY OUTCOMES:
procedure assesment | 1 month, 3 months, 6 months and 12 months
  By using:
  - VAS (ranging from 0: "No pain" to 100: "Maximum pain imaginable")
Assessing attention and working memory | 3 months and 12 months
  By using:
  - Trail Making Test (Reitan RM 1958) (2 parts A and B measured in seconds: The maximum score for part A is 100", 101" indicating that the test was not completed. The maximum score for Part B is 300", 301" indicating that the test was not completed)
qualitatively evaluate the effectiveness of the procedure | 3 months
  Semi-structured interviews with patients and their families oriented towards the evaluation of attention, affectivity and emotions.
Medication use | 1 month, 3 months, 6 months and 12 months
  Medication quantification scale (MQS) (Harden RN 2005): ranging from 0 (no antalgic medication used) to 126 (maximum antalgic medication used)
procedure assesment | 1 month, 3 months, 6 months and 12 months
  By using:
  - Hospital Anxiety and Depression scale (HAD) (Mykletun A 2001) (2 columns ranging from 0 " no or few anxiety" to 21 "high anxiety"
procedure assesment | 1 month, 3 months, 6 months and 12 months
  By using:
  - Global Perceived Effect scale (GPE, Kamper SJ 2010) (ranging from 1 "very bad" to 7 "very good")
Assessing attention and working memory | 3 months and 12 months
  By using:
  - WAIS-IV (Benson N 2010) ( 4 subtests submited with 10 items in all (ranging 0 to 19 each), to calculate intelligence quotient with a minimum at 0 and a maximum at 190)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul NGUYEN, Prof, Study Director — Clinique Bretéché ELSAN; Sylvain DURAND, Dr, Principal Investigator — Clinique Bretéché ELSAN
Locations (1):
- Clinique BRETECHE, Nantes, France

IPD SHARING:
Plan to Share IPD: No